CLINICAL TRIAL: NCT00066053
Title: Periodontal Intervention for Cardiac Events: A Pilot Trial
Brief Title: Periodontitis and Cardiovascular Events or "PAVE"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Robert J. Genco, DDS, PhD, Distinguished Professor, Vice Provost, STOR, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDCR-13940; U01DE013940 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2007-05

CONDITIONS: Cardiovascular Disease; Coronary Heart Disease; Myocardial Infarction; Cerebrovascular Accident
Keywords: Heart attacks; Stroke; Angina
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Stroke; Angina Pectoris | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Periodontal Treatment: SRP (Experimental): Comprehensive scaling & root planing and subgingival tissue removal; fluorides applied as appropriate; oral hygiene instructions.
  Interventions: Procedure: Periodontal Treatment: SRP
- Community Comparator (Active Comparator): Referral to community dentist with copy of x-rays and letter with diagnosis and recomendations for treatment.
  Interventions: Procedure: Referral

INTERVENTIONS:
Procedure: Periodontal Treatment: SRP — Scaling and root planing. Subgingival tissue removal. Fluorides as needed. Oral hygiene instructions. Oral hygiene instructions.
  Other Names: Treatment of periodontal infections.
  Arms: Periodontal Treatment: SRP
Procedure: Referral
  Arms: Community Comparator

SUMMARY:
The purpose of this study is to determine if treating periodontal infections (gum problems) will lead to fewer heart problems in patients at high risk for cardiovascular disease.

DETAILED DESCRIPTION:
There is growing evidence of a strong association between infection and atherosclerosis as well as a specific link between periodontal infection (gum problems) and heart disease. Previous studies have established possible effective treatments of periodontal disease. These treatments may lead to fewer heart events in persons at high risk for cardiovascular disease. In contrast to previous heart disease studies, the primary treatment in this project is directed toward infectious agents at periodontal sites. This project is a pilot randomized clinical trial to test the feasibility of selecting and refining a periodontal infection treatment and examining the effect of that treatment on future heart events. It is a multi-center planning and pilot study involving five investigational centers at the University at Buffalo (lead and overall coordinating center), University of North Carolina, Boston University, Kaiser Permanente/Oregon Health Science University, University of Maryland, and a data coordinating center at the University of North Carolina. Central microbiology and cytokine laboratories and a biologic specimen bank are also included. A team of cardiologists, periodontists, epidemiologists, infectious disease specialists, biostatisticians, research nurses in periodontics and cardiology, and data managers has been assembled to accomplish the research with a careful, cost-effective approach. The ultimate goal is to develop a definitive randomized clinical trial that will include about 4,000 participants from approximately 15 centers across the United States

ELIGIBILITY:
Eligibility:

* Aged 75 years or less AND 50% or more blockage of at least one artery in the heart,
* Heart problems in the last 3 years (including previous heart attack),
* Previous heart bypass surgery, or previous heart angioplasty with or without a stent, AND at least 6 natural teeth present in the mouth AND evidence of mild to severe gum problems.

Exclusion:

Any of the following:

* A major illness requiring hospitalization,
* Renal dialysis,
* Serum creatinine > 3 mg/dl,
* Organ transplant recipient requiring immunosuppression medication,
* Surgery needed in the next 3 years,
* Chemotherapy in the past 3 years,
* Head and/or neck radiation at any time in the past,
* Liver dysfunction,
* Class IV congestive heart failure,
* Drug or alcohol abuse,
* Pacemaker or AICD/defibrillator.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2003-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Patient outcomes are hospitalized for myocardial infarction (MI), cardiac revascularization, fatal coronary heart disease, unstable angina, and/or hospitalized ischemic stroke. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Sara G Grossi, DDS, MS, Principal Investigator — University at Buffalo; Thomas E van Dyke, DDS,MS, Principal Investigator — Goldman School of Dental Medicine, Boston, MA; John C Gunsolley, DDS,MS, Principal Investigator — University of Maryland, Dept. of Periodontics, Baltimore, MD; James D Beck, Ph.D, Principal Investigator — University of NC, School of Dentistry, Chapel Hill, NC; Lloyd E Chambless, PhD,, Principal Investigator — University of NC, Dept. of Biostatistics, Chapel Hill, NC; Steven Offenbacher, DDS,PhD,MMSc, Principal Investigator — University of NC, Comprehensive Cntr. for Inflammatory Diseases, Chapel Hill, NC; Theresa Madden, DDS, PhD, Principal Investigator — Oregon Health and Science University, Portland, OR; Gerardo Maupome, PhD, Principal Investigator — Kaiser-Permanente Center for Health Research, Portland, OR
Locations (1):
- University at Buffalo, Buffalo, New York, United States